CLINICAL TRIAL: NCT06151249
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study to Evaluate the Safety and Ability of Meritup Oral Liquid to Reduce Fatigue in Patients With Metastatic Breast Cancer Receiving Chemotherapy
Brief Title: Evaluate the Meritup Oral Solution to Decrease Fatigue in Metastatic Breast Cancer Patients Receiving Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chung Shan Medical University (Other)
Collaborators: Phytofound Biotech Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSMUH No:CS2-23089
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Fatigue
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Intervention Model Description: An add-on study design to assess the superiority of Meritup over placebo will be utilized in this study to evaluate whether Meritup can decrease fatigue in patients with fatigue. The study will be conducted as a double-blind, randomized trial.
Who Masked: Participant
Masking Description: Chemotherapy+Meritup Chemotherapy+Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy+Meritup (Experimental): Chemotherapy+Meritup 20ml TID
  Interventions: Combination Product: Meritup oral solution
- Chemotherapy+Placebo (Placebo Comparator): Chemotherapy+Placebo 20ml TID
  Interventions: Combination Product: Meritup oral solution

INTERVENTIONS:
Combination Product: Meritup oral solution — chemotherapy + Meritup

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel study to evaluate the safety profile and ability of Meritup oral solution to decrease fatigue in metastatic breast cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
The study population designed to be enrolled is patients with histologically and/or cytologically confirmed breast cancer with clinical evidence of recurrent or progressive metastatic disease and at least completed 3 cycle chemotherapy regimen who have evidence of fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients over 20years old and under 80 years old.
2. Estrogen receptor (ER), progesterone receptor (PR) and human epidermal growth factor receptor (HER2), These 3 indicators are all negative.
3. After at least 3 cycles of chemotherapy.
4. Sign the subject Informed Consent Form (ICF).

Exclusion Criteria:

1. Have received other clinical studies within 3 weeks
2. Any uncontrollable infection
3. History of lupus erythematosus, rheumatoid arthritis, ankylosing spondylosis, scleroderma or multiple sclerosis
4. History of cancer cells that have metastasized to the brain
5. Currently receiving a mixture of three or more types of cytotoxic chemotherapy drugs
6. Currently using anti-fatigue treatments, including psychostimulants, acupuncture, etc. Note: Antidepressants are used for treatment to relieve fatigue (such as depression or hot flashes) is allowed,
7. Need to use long-acting sustained-release pain narcotic analgesics
8. Uncontrollable nausea, vomiting or other symptoms that will hinder the ability to speak about the test product
9. Any other serious illness/history that would limit the patient's ability to receive study treatment, as determined by the researcher evaluate
10. Lactation, pregnancy or planning pregnancy
11. People with cardiovascular disease or severe liver and kidney dysfunction should not drink it within one week after surgery.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in fatigue scores | one months
  Changes in fatigue scores using the Functional Assessment of Chronic Illness Treatment (FACIT)-Fatigue subscale after 9 weeks of combined chemotherapy treatment

SECONDARY OUTCOMES:
Blood test | one month
  WBC, RBC, PLT, serum creatinine (SCr), SGOT, SGPT

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Hsin Yeh, MD, PhD, Principal Investigator — Chung Shan Medical University

IPD SHARING:
Plan to Share IPD: No